CLINICAL TRIAL: NCT05434793
Title: China Medical University, Taichung, Taiwan,
Brief Title: The Effect of Laser Acupuncture Stimuli at ZUSANLI(ST36) on Pulse Spectrum Variations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: /CMUH107-REC2-145
Record Dates: First submitted 2021-04-21; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Harmonic Wave
Keywords: Sham Acupuncture; Arterial Pulse; Fourier Transformation; Harmonics

STUDY DESIGN:
Intervention Model Description: In this study, the effects of sham acupuncture at Tsu San Li (St-36) were examined by analyzing noninvasive 30-sec. recordings of the radial arterial pulses for 3 groups of patients treated with different probes (blunt, sharp, and patch) on the superficial skin of the acupuncture point. The 3 groups were then treated with the sharp probe for 3 different periods (16, 30, and 50 seconds). Then the investigators compared the harmonics of the radial arterial pulse after Fourier transformation before and after the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The meridian effect of sham testing from mechanical stimulation (Experimental): The effects of sham acupuncture at Tsu San Li (St-36) were examined by analyzing noninvasive 30-sec. recordings of the radial arterial pulses for 3 groups of patients treated with different probes (blunt, sharp, and patch) on the superficial skin of the acupuncture point. The 3 groups were then treated with the sharp probe for 3 different periods (16, 30, and 50 seconds). Then we compared the harmonics of the radial arterial pulse after Fourier transformation before and after the treatment.
  Interventions: Device: RJ-LASER, LASERPEN®; Reimers & Janssen, Germany

INTERVENTIONS:
Device: RJ-LASER, LASERPEN®; Reimers & Janssen, Germany — The device was frequently used in laser acupuncture on the superficial skin of the acupuncture point Tsu San Li (St-36).

SUMMARY:
Background: Acupuncture has been criticized as a theatrical placebo for the sham effect. Unfortunately, sham tests used in control groups in acupuncture studies have always ignored the underlying biophysical factors, including resonance involved in acupuncture points and meridians.

Methods: In this study, the effects of sham acupuncture at Tsu San Li (St-36) were examined by analyzing noninvasive 30-sec. recordings of the radial arterial pulses for 3 groups of patients treated with different probes (blunt, sharp, and patch) on the superficial skin of the acupuncture point. The 3 groups were then treated with the sharp probe for 3 different periods (16, 30, and 50 seconds). Then the investigators compared the harmonics of the radial arterial pulse after Fourier transformation before and after the treatment.

DETAILED DESCRIPTION:
Acupuncture has been criticized as a theatrical placebo for its sham effect. It is unfortunate that sham tests designed as the control group in acupuncture studies have always ignored the biophysical factors, resonance, in acupuncture points, and thus have led to confusing results. The investigators' previous studies revealed that specific frequency effects are found at the acupuncture points on the Fourier components of the radial arterial pulse. The nearby non-acupuncture point also has similar but insignificant effects as the acupuncture point.

Meridians are the groups of acupuncture points, and can be measured from the harmonics of the arterial pulse, and thus physicians who practice traditional Chinese Medicine use the pulse to diagnose disease, to evaluate patients' physical conditions, and even to predict death. The importance of the information within arterial pulse waves has long been recognized in clinical medicine. Arterial pulse wave analysis has been widely used in clinical practice, for example, in cases of hypertension, cardiac failure, and aging. The investigators' previous studies revealed that the pulse spectrum of the radial arterial pulse could be highly correlated among patients with abnormal liver function. The specific Fourier components in the pulse provide more physiologic information than do systolic and diastolic blood pressure measurements during the process of dying. In addition, pulse spectrum analysis can be used to differentiate atopic dermatitis with the third harmonic of the radial pulse, and the fourth harmonic of the radial pulse wave has been shown to predict adverse cardiac events in asymptomatic patients with type 2 diabetes. Recently, pulse spectrum analysis has facilitated the diagnosis of coronary artery disease. The investigators can qualitatively and quantitatively gain physiologic or pathologic information by measuring the harmonics of blood pressure because the resonance in the cardiovascular system is highly efficient for hemodynamic evolution design. Each organ and its related meridian are in resonance with a specific Fourier component of pressure waves.

Meridians present in harmonics are the biophysical design for resonance, showing that the heart drives the cardiovascular system with less than 2 watts. This tiny factor, including acupuncture, moxibustion, massage, bian stone, and acupressure, which change resonance, will redistribute the hemodynamics of the cardiovascular system and then appear in the harmonics of the arterial pulse. If the investigators do not consider resonance, meridian, and acupuncture, the investigators will miss the effect when designing a sham test.

This study was derived from the sham test for laser acupuncture, and the results showed that the sham effect cannot be ignored. Thus, the investigators examined the effect of sham acupuncture at Tsu San Li (St-36) by noninvasively recording the radial arterial pulses for patients treated with different types of probes (blunt, sharp, and patch) on the superficial skin of the acupuncture point for 30 sec. A second group of patients was tested with a sharp probe for differing amounts of time (16, 30, and 50 sec.). The investigators then compared the harmonics of the radial arterial pulse after the Fourier transformation before and after the treatment. The investigators hypothesized that harmonics could be physiologic indicators corresponding with the resonance on the tiny change of acupuncture point, and could explain the sham effect found in clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* OPD patients

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
The Magnitude Value of Harmonic Effects of Sham Acupuncture at Tsu San Li (St-36) in the Radial Pulse Wave | two-year study
The Phase Value of Harmonic Effects of Sham Acupuncture at Tsu San Li (St-36) in the Radial Pulse Wave | two-year study

CONTACTS AND LOCATIONS:
Locations (1):
- Yu- Cheng Kuo, Taipei, Taiwan